CLINICAL TRIAL: NCT02368405
Title: Nutrition Education for Cardiovascular Disease Prevention in Individuals With Spinal Cord Injury
Brief Title: Nutrition Education for Cardiovascular Disease Prevention in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 09-14-06E
Record Dates: First submitted 2015-02-10; First posted 2015-02-23 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study allocation was placed in concealed envelopes by research volunteer who was not otherwise involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Control group will receive standard of care
  Interventions: Behavioral: Control
- Treatment (Experimental): Participants in the treatment group will receive six interactive nutrition lectures over the course of three weeks. The treatment program is titled "Eat Smart, Live Better"
  Interventions: Behavioral: Eat Smart, Live Better

INTERVENTIONS:
Behavioral: Control — Participants in the control group will receive the standard nutrition lecture currently given at Carolinas Rehabilitation to all inpatients with spinal cord injuries. This one lecture is what is required by Commission on Accreditation for Rehabilitation Facilities (CARF)
  Arms: Control
Behavioral: Eat Smart, Live Better — Intervention participants will participate in a series of six, 60-minute small group sessions of interactive nutrition education discussions led by a Registered Dietitian delivered over 3 weeks. They will also have one follow-up comprehensive nutrition education session approximately 3 months after receipt of the Eat Smart, Live Better curriculum. In order to help us assess the effectiveness of the nutrition education program, we will assess nutrition behavior and knowledge at this time as well. Community participants in the treatment group will attend the sessions at Carolinas Rehabilitation (CR). The control participants from the community will come to CR for the one standard nutrition lecture. Caregivers and spouses of all of the participants will be encouraged to attend the sessions.
  Arms: Treatment

SUMMARY:
This is a randomized controlled trial to study a nutrition education intervention in individuals with spinal cord injuries both in the acute rehabilitation setting (n = 100) and the community setting (n = 100). Participants in the treatment group will receive six interactive nutrition lectures based upon a successful program that has been used in older adults titled "Eat Smart, Stay Well". The goals of intervention are to improve whole-grain, fruit and vegetable, and low-fat dairy intake and reduce fat and saturated fat intake. Secondary outcomes will include improvements in waist circumference of body mass index and some biomarkers such as cholesterol and blood sugar.

DETAILED DESCRIPTION:
The prevalence of SCI is significant. Obesity, diabetes, and CVD are more prevalent in the SCI population. Many individuals with SCI are unable or have a limited capacity to exercise. This reality makes good nutrition even more urgent. This study will be the first to test whether additional nutrition education can improve nutrition behavior and knowledge, diet quality, adiposity, and metabolic CVD risk factors in individuals with SCI and to determine the best setting to deliver nutrition education to individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Injury Association classification A, B, C as long as they are not functional ambulators

Exclusion Criteria:

* Stage III or IV pressure ulcers, pregnancy, end-stage renal disease, treatment for cancer except for nonmelanoma skin cancer within the past five years, and chronic, nontobacco substance-abuse, cognitive impairment with inability to learn

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Nutrition Behavior and Knowledge, measured by Likert scale | Change from baseline at three months, and 12 months
  Nutrition behavior will be recorded from two five point Likert scale questions ranging from 1 = not practicing the behavior to 5 = practicing it regularly. Questions are related to eating fruits and vegetables and to decreasing fat intake. The recorded scores for these questions will be pooled for nutrition behavior and range from 2 = very low to 10 = very high.

SECONDARY OUTCOMES:
Body Mass Index | Baseline and 12 months
  participants will be weighed and measured and BMI calculated
Waist Circumference | Baseline and 12 months
Laboratories - Fasting lipid panel | Baseline and 12 months
  Fasting lipid panel
Laboratories - Fasting blood glucose | Baseline and 12 months
  Fasting blood glucose
Laboratories - High Sensitivity C-reactive protein | Baseline and 12 months
  High Sensitivity C-reactive protein
Diet quality as measured by Diet History Questionnaire (DHQ) II | Baseline and 12 months
  The Diet History Questionnaire (DHQ) II will be administered. Each participant will be assessed for fruit, vegetable, dairy, whole-grain, lean protein, fat, and saturated fat intake. Intake for each food group will also be checked for compliance with the 2010 Dietary Guidelines for Americans.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse A Lieberman, MD, MSPH, Principal Investigator — Carolinas Rehabilitation
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hooper L, Abdelhamid AS, Jimoh OF, Bunn D, Skeaff CM. Effects of total fat intake on body fatness in adults. Cochrane Database Syst Rev. 2020 Jun 1;6(6):CD013636. doi: 10.1002/14651858.CD013636. PMID 32476140
- [Derived] Lieberman JA, McClelland JW, Goff DC Jr, Racine E, Dulin MF, Bauman WA, Niemeier J, Hirsch MA, Norton HJ, Moore CG. Nutrition education for cardiovascular disease prevention in individuals with spinal cord injuries: study protocol for a randomized controlled trial. Trials. 2017 Dec 4;18(1):584. doi: 10.1186/s13063-017-2263-2. PMID 29202852

DOCUMENTS (1):
  • Informed Consent Form (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT02368405/ICF_000.pdf